CLINICAL TRIAL: NCT01830140
Title: A Safety Study of Bimatoprost in Patients With Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 192024-081
Record Dates: First submitted 2013-04-10; First posted 2013-04-12 (Estimated); Results first posted 2015-05-06 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-04

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bimatoprost 0.01% (Experimental): Bimatoprost 0.01% (LUMIGAN® 0.01%) administered each evening in both eyes for 6 weeks.
  Interventions: Drug: Bimatoprost 0.01%
- Bimatoprost 0.03% (Active Comparator): Bimatoprost 0.03% (LUMIGAN® 0.03%) administered each evening in both eyes for 6 weeks.
  Interventions: Drug: Bimatoprost 0.03%

INTERVENTIONS:
Drug: Bimatoprost 0.01% — Bimatoprost 0.01% (LUMIGAN® 0.01%) administered each evening in both eyes for 6 weeks.
  Other Names: LUMIGAN® 0.01%
  Arms: Bimatoprost 0.01%
Drug: Bimatoprost 0.03% — Bimatoprost 0.03% (LUMIGAN® 0.03%) administered each evening in both eyes for 6 weeks.
  Other Names: LUMIGAN® 0.03%
  Arms: Bimatoprost 0.03%

SUMMARY:
This safety study will evaluate bimatoprost 0.01% and 0.03% in patients with glaucoma or ocular hypertension (OHT).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of glaucoma or ocular hypertension

Exclusion Criteria:

* Active ocular disease other than glaucoma or ocular hypertension
* Require chronic use of ocular medications other than the study medication during the study (intermittent use of artificial tear solution will be permitted)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 466 (Actual)
Dates: Start 2013-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (2):
- United States (2):
  - Artesia, California
  - El Paso, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bimatoprost 0.01% | Bimatoprost 0.03%
Started | 233 | 233
Completed | 226 | 229
Not Completed | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bimatoprost 0.01% | Bimatoprost 0.03% | Total
Number analyzed (Participants) | 233 | 233 | 466
Age, Customized [Number; unit: Participants]
  < 45 years | 6 | 7 | 13
  Between 45 and 65 years | 91 | 97 | 188
  ≥65 years | 136 | 129 | 265
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 158 | 299
  Male | 92 | 75 | 167

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With an Increase in Macroscopic Conjunctival Hyperemia in Either Eye
Description: Macroscopic conjunctival hyperemia (eye redness) is graded in each eye on a 5-point scale (Scale 0 to +3: none, trace, mild, moderate, severe). An increase (worsening) in macroscopic conjunctival hyperemia is defined as an increase in macroscopic conjunctival hyperemia grade of at least 1 from baseline in either eye.
Time Frame: Baseline, 6 Weeks
Population: Intent-to-Treat: all randomized patients
Measure: Number; unit: Percentage of Patients
Arm/Group | Bimatoprost 0.01% | Bimatoprost 0.03%
Number analyzed (Participants) | 233 | 233
Percentage of Patients | 34.3 | 39.1

ADVERSE EVENTS:
Arm/Group | Bimatoprost 0.01% | Bimatoprost 0.03%
Serious Adverse Events (participants affected / at risk) | 2/233 | 2/233
Other Adverse Events (participants affected / at risk) | 49/233 | 66/233
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Bimatoprost 0.01% (N=233) | Bimatoprost 0.03% (N=233)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 0
Monoplegia (Nervous system disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/92 | 1/75
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost 0.01% (N=233) | Bimatoprost 0.03% (N=233)
Eye Pruritus (Eye disorders) | 7 | 13
Conjunctival Hyperaemia (Eye disorders) | 42 | 53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.